CLINICAL TRIAL: NCT07390604
Title: Case Series : Management of Elevated Lipoprotein(a) Using Double-Filtration Plasmapheresis (DFPP) in Hemodialysis Patients With Chronic Kidney Disease Clinical and Biological Outcomes in Patients at Cardiovascular and Thromboembolic Risk
Brief Title: Case Series : Management of Elevated Lipoprotein(a) Using Double-Filtration Plasmapheresis (DFPP) in Hemodialysis Patients With Chronic Kidney Disease ; ( LiPo-A )
Acronym: LiPo-A
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-03Obs-CHRMT
Record Dates: First submitted 2026-01-14; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lipoprotein(a); Lipoprotein-apheresis; Double-filtration Plasmapheresis; Hemodialysis Complication; End Stage Chronic Renal Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lipoprotein-apheresis DFPP has been performed in patients with Lp(a) levels greater than 125 nmol/L. In this report, data will be presented on five hemodialysis patients with significantly elevated Lp(a) levels (>200 nmol/L) who had a history of cardiovascular disease and notable thromboembolic events.

DETAILED DESCRIPTION:
The biological and clinical outcomes related to Lipoprotein-apheresis DFPP treatment and the associated cardiovascular and thromboembolic events will be described in these patients. Additionally, the impact of DFPP on biological and clinical markers including LDL cholesterol, triglycerides, fibrinogen, hemoglobin, platelet count, C-reactive protein (CRP), blood pressure, plasma volume treated, volume of albumin substitution, volume of plasma rejected, and duration of each Lipoprotein-apheresis DFPP session will be evaluated .

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients with elevated Lp(a) levels (>200 nmol/L) and a history of cardiovascular disease and/or thromboembolic events who underwent DFPP sessions as part of their management

Exclusion Criteria:

* -Patients with progressive, active disease, presenting with severe general deterioration and a limited life expectancy
* Patients presenting with hemodynamic instability
* Patients presenting with acute kidney diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: chronic Hemodialsisi patients
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
serum Lp(a) concentration (nmol/L), on routine venous blood sampling | up to 15 months after inclusion
  Before and after each DFPP session (repeated measures) during the study period

SECONDARY OUTCOMES:
serum LDL and serum triglycerides concentration (g/L), on routine venous blood sampling | up to 15 months after inclusion
  before and after each DFPP session (repeated measures) during the study period
serum triglycerides concentration (g/L), on routine venous blood sampling | up to 15 months after inclusion
  before and after each DFPP session (repeated measures) during the study period
cardiovascular or thromboembolic events | during all the study period: up to 15 months after inclusion
  Myocardial infarction, stroke, Deep vein thrombosis, Pulmonary embolism, Systemic arterial embolism, aortiques complictions, thrombosis, Based on patient questioning and clinical examination during routine follow-up consultations
Hemodynamic status:blood pressure | up to 15 months after inclusion
  follow-up of patients' blood pressure (mmHg) before and after each DFPP session (repeated measures) during the study period
Hemodynamic status: ultrafiltration rate | up to 15 months after inclusion
  follow-up of patients' ultrafiltration rate (grams) before and after each DFPP session (repeated measures) during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Zead TUBAIL, MD, Principal Investigator — CHR Metz-Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No